CLINICAL TRIAL: NCT03743766
Title: A Phase II Study of Anti-PD1 Monoclonal Antibody (Nivolumab, BMS-936558) Administered in Combination with Anti-LAG3 Monoclonal Antibody (Relatlimab, BMS-986016) in Patients with Metastatic Melanoma Naïve to Prior Immunotherapy in the Metastatic Setting
Brief Title: Nivolumab, BMS-936558 in Combination with Relatlimab, BMS-986016 in Patients with Metastatic Melanoma Naïve to Prior Immunotherapy in the Metastatic Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Kirkwood (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, John Kirkwood, Usher Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-071
Record Dates: First submitted 2018-10-18; First posted 2018-11-16 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Melanoma
Keywords: Stage IIIB; Stage IIIC; Stage IIID; Stage IV; immune checkpoint blockade (ICB); Lymphocyte activation gene-3 (LAG3; CD223); immunotherapy
MeSH Terms: conditions — Melanoma | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Intervention Model Description: In the 4-week lead-in phase, subjects will be randomized to one of three arms for 1 cycle (4 weeks) of lead-in treatment with nivolumab, relatlimab, or the combination of nivolumab and relatlimab. Following 1 cycle of lead-in treatment, all subjects will be treated with the combination of relatlimab and nivolumab every 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Relatlimab (Experimental): Cycle 1: Relatlimab (BMS-986016) is supplied as a sterile 10mg/mL formulation to be administered as an intravenous (IV) infusion at 160 mg IV for the first 4 weeks (cycle 1).
  Cycle 2+: Combination therapy will be administered by sequential infusion. Nivolumab administered at 480 mg IV followed by infusion of relatlimab at 160 mg IV once every 4 weeks.
  Interventions: Drug: Relatlimab
- Nivolumab (Experimental): Cycle 1: Nivolumab (BMS-936558) is supplied as a sterile 10-mg/mL formulation to be administered as an IV infusion at 480 mg IV for the first 4 weeks.
  Cycle 2+: Combination therapy will be administered by sequential infusion. Nivolumab administered at 480 mg IV followed by infusion of relatlimab at 160 mg IV once every 4 weeks.
  Interventions: Drug: Nivolumab
- Relatlimab + Nivolumab (Experimental): Cycle 1+: Combination therapy will be administered by sequential infusion. Nivolumab administered at 480 mg IV followed by infusion of relatlimab at 160 mg IV for the first 4 weeks (Cycle 1), then once every 4 weeks afterwards.
  Interventions: Drug: Relatlimab + Nivolumab

INTERVENTIONS:
Drug: Relatlimab — Relatlimab (BMS-986016) - 10mg/mL formulation to be administered as an intravenous (IV) infusion at 160 mg IV.
  Other Names: BMS-986016
  Arms: Relatlimab
Drug: Nivolumab — Nivolumab (BMS-936558) - 10-mg/mL formulation to be administered as an IV infusion at 480 mg IV.
  Other Names: BMS-936558
  Arms: Nivolumab
Drug: Relatlimab + Nivolumab — Combination (Relatlimab + Nivolumab) therapy will be administered by sequential infusion. Nivolumab administered at 480 mg IV followed by infusion of relatlimab at 160 mg IV.
  Other Names: BMS-986016 and BMS-936558
  Arms: Relatlimab + Nivolumab

SUMMARY:
The main goal of this study is to evaluate the antitumor activity of relatlimab and nivolumab in combination in subjects with unresectable or metastatic melanoma who have not received prior treatment with immunotherapy.

DETAILED DESCRIPTION:
This study will evaluate the antitumor activity of anti-LAG3 monoclonal antibody relatlimab and the anti-PD1 monoclonal antibody nivolumab in combination in subjects with unresectable or metastatic melanoma who have not received prior treatment with immunotherapy. The trial is designed with a lead-in phase of 2 cycles (4 week) treatment of either nivolumab, relatlimab, or the combination of nivolumab/relatlimab, followed by a combination phase of nivolumab/relatlimab treatment in all subjects. This lead-in design with accompanying tumor biopsies and peripheral blood analyses will enable mechanistic analyses of the effect of LAG3 and PD1 blockade alone and in combination to enhance understanding of mechanisms of response and resistance. Duration of response, progression free survival, and safety will be assessed as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

• Men or women 18 years of age or older meeting AJCC 8th edition criteria for unresectable stage IIIB, stage IIIC, stage IIID, or stage IV melanoma who have not received treatment with immunotherapy in the metastatic setting

Exclusion Criteria:

* Known or suspected CNS metastases, with the following exceptions:

  * Subjects with controlled brain metastases will be allowed to enroll. Controlled brain metastases are defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment at the time of consent. Subjects must be off steroids for at least 2 weeks prior to randomization.
  * Subjects with signs or symptoms of brain metastases are not eligible unless brain metastases are ruled out by computed tomography or magnetic resonance imaging.
* Active autoimmune disease requiring treatment, with the exception of type 1 diabetes mellitus, vitiligo, resolved childhood asthma/atopy, controlled hyper/hypothyroidism, hypoadrenalism or hypopituitarism.
* Prior systemic treatment in the metastatic setting, including anti-PD1, anti-PDL1, anti-PDL2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways; or chemotherapy.
* Prior adjuvant treatment with anti-PD1, anti-PDL1, and/or anti-LAG3 antibody. Note that prior adjuvant treatment with targeted therapy (e.g. BRAF/MEK inhibition), anti-CTLA4, or treatment not otherwise specified above would be permitted.
* Ocular melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Change in LAG3 Expression | At baseline and at 4 weeks
  LAG3 (cell surface molecule expressed on activated T cells) expression is either positive (present) or not detectable if absent after completion of lead-in phase.
Change in PD1 expression | At baseline and at 4 weeks
  PD1 (programmed cell death protein 1) expression is either positive (present) or not detectable if absent after completion of lead-in phase
Change in Tumor Size | At baseline and at 4 weeks
  Tumor size will be assessed per Response Evaluation Criteria in Solid Tumors. Per RECIST 1.1, Tumour lesions: Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:
  * 10 mm by CT scan (CT scan slice thickness no greater than 5 mm; see Appendix II on imaging guidance).
  * 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable).
  * 20 mm by chest X-ray.
Overall Response Rate (ORR) | Beginning at 12 weeks post initial treatment, up to 4 years
  Number of participants experiencing Complete Response (CR) + Number of participants experiencing Partial Response (PR)/total patients assessed. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

SECONDARY OUTCOMES:
Clinical Benefit Rate | 12 weeks post initial treatment, up to 4 years
  Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) / total patients assessed per RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Duration of Response | 12 weeks post initial treatment, up to 4 years
  Time from first documented Complete Response (CR) or Partial Response (PR) until the first date that progressive disease is objectively documented. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free Survival (PFS) | Up to 4 years
  Progression-free survival is defined as the time between the date of randomization and the first date of documented progression or death due to any cause, whichever occurs first. Per RECIST v1.1, Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Overall Survival (OS) | Up to 4 years
  Overall survival is defined as the time between the date of randomization and the date of death due to any cause.
LAG3 Expression | At week 16 (2 weeks post combination treatment (3 cycles))
  LAG3 (cell surface molecule expressed on activated T cells) expression (positive (present) or not detectable if absent) in tumor and peripheral blood of treated participants who experience a complete response, partial response, or stable disease, prior to ultimately experiencing disease progression.
PD-1 Expression | At week 16 (12 weeks post combination treatment (3 cycles))
  PD-1 (programmed cell death protein 1) expression (positive (present) or not detectable if absent) in tumor and peripheral blood of treated participants who experience a complete response, partial response, or stable disease, prior to ultimately experiencing disease progression.
Change in CD4+ tumor infiltrating lymphocytes | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Percentage and number of CD4+ tumor infiltrating lymphocytes present
Change in CD8+ tumor infiltrating lymphocytes | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Percentage and number of CD8+ tumor infiltrating lymphocytes present
Change in granzyme B serum levels | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Level of granzyme B (a serine protease secreted cells to mediate apoptosis in target cells) in serum.
Change in cell effector/memory status | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Measure of cells that have previously encountered and responded to their cognate antigen.
Change in activation and maturation of dendritic cells | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Measure of expression of activation and maturation of dendritic cells
Change in T cell count | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Number of T cells present in blood and tumor
Change in T cell count | At the time of disease progression - up to 4 years
  Number of T cells present in blood and tumor in patients that had previously demonstrated complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Change in soluble LAG3 levels | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Amount of LAG3 (cell surface molecule expressed on activated T cells) protein present in blood and tumor tissue.
Soluble LAG3 levels | At the time of disease progression - up to 4 years
  Amount of LAG3 (cell surface molecule expressed on activated T cells) protein present in blood and tumor tissue in patients that had previously demonstrated complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Change in Regulatory T cell (Treg) marker level | At 2 weeks prior first study treatment, at 4 weeks, at 12 weeks
  Amount of Regulatory T cell (Treg) markers present in blood and tumor tissue.
Regulatory T cell (Treg) marker levels | At the time of disease progression - up to 4 years
  Amount of Regulatory T cell (Treg) markers present in blood and tumor tissue.in patients that had previously demonstrated complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

OTHER OUTCOMES:
Single cell RNA sequencing | 2 weeks
  The presence and quantity of RNA in in blood and tumor tissue.
Single cell RNA sequencing | At 4 weeks post Cycle 1
  The presence and quantity of RNA in in blood and tumor tissue.
Single cell RNA sequencing | At week 16 (12 weeks post combination treatment (3 cycles)
  The presence and quantity of RNA in in blood and tumor tissue.
Single cell RNA sequencing | At the time of disease progression - up to 4 years
  The presence and quantity of RNA in in blood and tumor tissue in patients that had previously demonstrated complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkwood, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No